CLINICAL TRIAL: NCT03120013
Title: Rehabilitative Trial With Cerebello-Spinal tDCS for the Treatment of Neurodegenerative Ataxia
Brief Title: Rehabilitative Trial With Cerebello-Spinal tDCS in Neurodegenerative Ataxia
Acronym: CStDCSAtaxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Barbara Borroni, Professor, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NP1576
Record Dates: First submitted 2017-04-14; First posted 2017-04-19 (Actual); Results first posted 2019-06-28 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Ataxia, Cerebellar; Cerebellar Ataxia; Spinocerebellar Ataxias; Ataxia, Spinocerebellar; Spinocerebellar Ataxia Type 1; Spinocerebellar Ataxia Type 2; Spinocerebellar Ataxia 3; Spinocerebellar Degenerations; Friedreich Ataxia; Ataxia With Oculomotor Apraxia; Multiple System Atrophy
Keywords: Transcranial direct current stimulation; Transcranial magnetic stimulation; Spinocerebellar ataxia; Cerebellar ataxia
MeSH Terms: conditions — Cerebellar Ataxia; Spinocerebellar Ataxias; Machado-Joseph Disease; Spinocerebellar Degenerations; Friedreich Ataxia; Spinocerebellar ataxia, autosomal recessive 1; Multiple System Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Real tDCS (Experimental): 10 days anodal cerebellar and cathodal spinal tDCS
  Interventions: Device: Anodal cerebellar and cathodal spinal tDCS
- Sham tDCS (Sham Comparator): 10 days sham cerebellar and sham spinal tDCS
  Interventions: Device: Sham cerebellar and sham spinal tDCS

INTERVENTIONS:
Device: Anodal cerebellar and cathodal spinal tDCS — 10 sessions of anodal cerebellar and cathodal spinal transcranial direct current stimulation (5 days/week for 2 weeks)
  Arms: Real tDCS
Device: Sham cerebellar and sham spinal tDCS — 10 sessions of sham cerebellar and sham spinal transcranial direct current stimulation (5 days/week for 2 weeks)
  Arms: Sham tDCS

SUMMARY:
Neurodegenerative cerebellar ataxias represent a group of disabling disorders for which we currently lack effective therapies. Cerebellar transcranial direct current stimulation (tDCS) is a non-invasive technique, which has been demonstrated to modulate cerebellar excitability and improve symptoms in patients with cerebellar ataxias. In this randomized, double-blind, sham-controlled study, the investigators will evaluate whether a two-weeks' treatment with cerebellar anodal tDCS and spinal cathodal tDCS can improve symptoms in patients with neurodegenerative cerebellar ataxia and can modulate cerebello-motor connectivity, at short and long term.

DETAILED DESCRIPTION:
Neurodegenerative cerebellar ataxias represent a heterogeneous group of disabling disorders in which progressive ataxia of gait, limb dysmetria, oculomotor deficits, dysarthria and kinetic tremor are the prominent clinical manifestations. Both the hereditary and sporadic forms usually present in young adulthood, and are characterized by atrophy of cerebellar or brainstem structures. Currently, cerebellar ataxia lack effective disease-modifying therapies.

Cerebellar transcranial direct current stimulation (tDCS) is a non-invasive technique, which has been demonstrated to modulate cerebellar excitability and improve symptoms in patients with cerebellar ataxias. The present randomized, double-blind, sham-controlled study will investigate whether a two-weeks' treatment with cerebellar anodal tDCS and spinal cathodal tDCS can improve symptoms in patients with neurodegenerative cerebellar ataxia and can modulate cerebello-motor connectivity, at short and long term.

Subjects will be randomized in two groups, one receiving a 10 day (5 days/week for 2 weeks) treatment with anodal cerebellar and cathodal spinal tDCS and the other receiving sham stimulation with identical parameters. After the intervention, patients will be reassessed with a clinical and neurophysiological evaluation at 2 weeks, 1 months and 3 month after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a cerebellar syndrome and quantifiable cerebellar atrophy

Exclusion Criteria:

* Severe head trauma in the past
* History of seizures
* History of ischemic stroke or hemorrhage
* Pacemaker
* Metal implants in the head/neck region
* Severe comorbidity
* Intake of illegal drugs
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Borroni, MD, Principal Investigator — Azienda Ospedaliera Spedali Civili, Brescia; Alberto Benussi, MD, Principal Investigator — Università degli Studi di Brescia
Locations (1):
- AO Spedali Civili, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benussi A, Koch G, Cotelli M, Padovani A, Borroni B. Cerebellar transcranial direct current stimulation in patients with ataxia: A double-blind, randomized, sham-controlled study. Mov Disord. 2015 Oct;30(12):1701-5. doi: 10.1002/mds.26356. Epub 2015 Aug 14. PMID 26274840
- [Background] Benussi A, Dell'Era V, Cotelli MS, Turla M, Casali C, Padovani A, Borroni B. Long term clinical and neurophysiological effects of cerebellar transcranial direct current stimulation in patients with neurodegenerative ataxia. Brain Stimul. 2017 Mar-Apr;10(2):242-250. doi: 10.1016/j.brs.2016.11.001. Epub 2016 Nov 3. PMID 27838276
- [Background] Bikson M, Grossman P, Thomas C, Zannou AL, Jiang J, Adnan T, Mourdoukoutas AP, Kronberg G, Truong D, Boggio P, Brunoni AR, Charvet L, Fregni F, Fritsch B, Gillick B, Hamilton RH, Hampstead BM, Jankord R, Kirton A, Knotkova H, Liebetanz D, Liu A, Loo C, Nitsche MA, Reis J, Richardson JD, Rotenberg A, Turkeltaub PE, Woods AJ. Safety of Transcranial Direct Current Stimulation: Evidence Based Update 2016. Brain Stimul. 2016 Sep-Oct;9(5):641-661. doi: 10.1016/j.brs.2016.06.004. Epub 2016 Jun 15. PMID 27372845
- [Background] Rossini PM, Burke D, Chen R, Cohen LG, Daskalakis Z, Di Iorio R, Di Lazzaro V, Ferreri F, Fitzgerald PB, George MS, Hallett M, Lefaucheur JP, Langguth B, Matsumoto H, Miniussi C, Nitsche MA, Pascual-Leone A, Paulus W, Rossi S, Rothwell JC, Siebner HR, Ugawa Y, Walsh V, Ziemann U. Non-invasive electrical and magnetic stimulation of the brain, spinal cord, roots and peripheral nerves: Basic principles and procedures for routine clinical and research application. An updated report from an I.F.C.N. Committee. Clin Neurophysiol. 2015 Jun;126(6):1071-1107. doi: 10.1016/j.clinph.2015.02.001. Epub 2015 Feb 10. PMID 25797650
- [Background] Miranda PC, Salvador R, Wenger C, Fernandes SR. Computational models of non-invasive brain and spinal cord stimulation. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:6457-6460. doi: 10.1109/EMBC.2016.7592207. PMID 28269725
- [Background] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Background] Fiocchi S, Ravazzani P, Priori A, Parazzini M. Cerebellar and Spinal Direct Current Stimulation in Children: Computational Modeling of the Induced Electric Field. Front Hum Neurosci. 2016 Oct 17;10:522. doi: 10.3389/fnhum.2016.00522. eCollection 2016. PMID 27799905
- [Background] van Dun K, Bodranghien F, Manto M, Marien P. Targeting the Cerebellum by Noninvasive Neurostimulation: a Review. Cerebellum. 2017 Jun;16(3):695-741. doi: 10.1007/s12311-016-0840-7. PMID 28032321
- [Result] Benussi A, Dell'Era V, Cantoni V, Bonetta E, Grasso R, Manenti R, Cotelli M, Padovani A, Borroni B. Cerebello-spinal tDCS in ataxia: A randomized, double-blind, sham-controlled, crossover trial. Neurology. 2018 Sep 18;91(12):e1090-e1101. doi: 10.1212/WNL.0000000000006210. Epub 2018 Aug 22. PMID 30135258

RESULTS

PARTICIPANT FLOW:
Groups:
- Real tDCS, Then Sham tDCS: Participants first received real tDCS (anodal cerebellar and cathodal spinal tDCS) 5 days/week for 2 weeks. After a washout period of 6 months, they then received sham tDCS (sham cerebellar and sham spinal tDCS) 5 days/week for 2 weeks.
- Sham tDCS, Then Real tDCS: Participants first received sham tDCS (sham cerebellar and sham spinal tDCS) 5 days/week for 2 weeks. After a washout period of 6 months, they then received real tDCS (anodal cerebellar and cathodal spinal tDCS) 5 days/week for 2 weeks.
Period: First Intervention (2 Weeks)
Arm/Group | Real tDCS, Then Sham tDCS | Sham tDCS, Then Real tDCS
Started | 10 | 11
Received Intervention | 10 | 11
Completed | 10 | 10
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout (6 Months)
Arm/Group | Real tDCS, Then Sham tDCS | Sham tDCS, Then Real tDCS
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention (2 Weeks)
Arm/Group | Real tDCS, Then Sham tDCS | Sham tDCS, Then Real tDCS
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis are reported for 20 participants who completed the first intervention
Groups:
- All Study Participants: Participants who were randomized to receive either real tDCS or sham tDCS
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 20
Scale for the Assessment and Rating of Ataxia (SARA) score [Mean (Standard Deviation); unit: units on a scale] — Scale for the Assessment and Rating of Ataxia (SARA): clinical scale that is based on a semi-quantitative assessment of cerebellar ataxia on an impairment level. It consists of an 8-item performance based scale, yielding a total score of 0 (no ataxia) to 40 (most severe ataxia).
  units on a scale | 20.2 (7.4)
International Cooperative Ataxia Rating Scale (ICARS) score [Mean (Standard Deviation); unit: units on a scale] — International Cooperative Ataxia Rating Scale (ICARS): semi-quantitative 100-point scale consisting of 19 items divided into 4 weighted subscores including posture and gait disturbances, limb kinetic function, speech disorder, and oculomotor deficits, yielding a total score of 0 (no ataxia) to 100 (most severe ataxia).
  units on a scale | 53.0 (18.6)
9 Hole Peg Test (Dominant hand) [Mean (Standard Deviation); unit: seconds] — 4 timed trials of the 9 hole peg test (9HPT) were performed and averaged (mean values are reported) for each separate hand (dominant and nondominant). The 9HPT is a commonly used test to assess finger dexterity: the patient picks the pegs 1 at time and puts them in 9 holes on a peg board until all holes are filled and then removes them 1 at a time as quickly as possible. The total time to complete the task is recorded for each trial and for each separate hand (dominant and nondominant). Longer times represent greater impairment.
  seconds | 53.0 (24.3)
9 Hole Peg Test (non-Dominant hand) [Mean (Standard Deviation); unit: seconds] — 4 timed trials of the 9 hole peg test (9HPT) were performed and averaged (mean values are reported) for each separate hand (dominant and nondominant). The 9HPT is a commonly used test to assess finger dexterity: the patient picks the pegs 1 at time and puts them in 9 holes on a peg board until all holes are filled and then removes them 1 at a time as quickly as possible. The total time to complete the task is recorded for each trial and for each separate hand (dominant and nondominant). Longer times represent greater impairment.
  seconds | 56.1 (21.5)
8 Meter Walking Time [Mean (Standard Deviation); unit: seconds] — 4 timed trials of the 8 meter walking time (8MW) were performed and averaged (mean values are reported). The 8MW is defined as the time needed to walk 8 m as quickly as possible but safely with any device but without the help of another person or wall. Longer times represent greater impairment.
  seconds | 9.4 (3.4)
Short-Form Health Survey 36 [Mean (Standard Deviation); unit: units on a scale] — The Italian version of the Short-Form Health Survey 36 (SF-36), an interview-administered self-reported scale consisting of 36 scaled scores assessing 8 subdomains (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health, communication, psychosocial and energy), was used to assess changes in the patient's quality of life. The scale ranges from 0 (more disability) to 100 (less disability).
  units on a scale | 54.7 (17.5)
Cerebellar Brain Inhibition [Mean (Standard Deviation); unit: milli volt] — Cerebellar brain inhibition (CBI) is evaluated with a transcranial magnetic stimulation (TMS) protocol, using two coils. One placed over the cerebellar hemisphere and the other positioned on the contralateral primary motor cortex, with motor evoked potentials (MEPs) recorded on the first dorsal interosseous muscle. CBI measures the inhibition exerted by cerebellar structures on the motor cortex, and thus on MEPs amplitude, reflecting the integrity of the cerebellar-thalamo-cortical pathway. Lower values reflect higher inhibition and thus reduced impairment.
  milli volt | 0.94 (0.12)

OUTCOME MEASURES:

1. Primary Outcome: Change in the International Cooperative Ataxia Rating Scale (ICARS) Score From Baseline
Description: International Cooperative Ataxia Rating Scale (ICARS): semi-quantitative 100-point scale, yielding a total score of 0 (no ataxia) to 100 (most severe ataxia).
Time Frame: Baseline - 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 53.0 (18.6) | 52.7 (19.4)
  2 Weeks | 43.0 (19.6) | 52.1 (19.7)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Superiority; p < 0.001, ANCOVA

2. Primary Outcome: Change in the Scale for the Assessment and Rating of Ataxia (SARA) Score From Baseline
Description: Scale for the Assessment and Rating of Ataxia (SARA): 8-item performance based scale, yielding a total score of 0 (no ataxia) to 40 (most severe ataxia).
Time Frame: Baseline - 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale | 15.8 (7.6) | 19.7 (7.5)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Superiority; p < 0.001, ANCOVA

3. Secondary Outcome: Change in the International Cooperative Ataxia Rating Scale (ICARS) Score From Baseline
Description: as for outcome 1
Time Frame: Baseline - 2 weeks - 1 month - 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 53.0 (18.6) | 52.7 (19.4)
  2 Weeks | 43.0 (19.6) | 52.1 (19.7)
  1 Month | 41.3 (19.6) | 52.5 (19.2)
  3 Months | 44.2 (19.6) | 52.4 (19.4)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Superiority; p < 0.001, ANCOVA

4. Secondary Outcome: Change in the Scale for the Assessment and Rating of Ataxia (SARA) Score From Baseline
Description: as for outcome 2
Time Frame: Baseline - 2 weeks - 1 month - 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 20.2 (7.3) | 19.9 (7.3)
  2 Weeks | 15.8 (7.6) | 19.7 (7.5)
  1 Month | 15.1 (7.7) | 19.7 (7.3)
  3 Months | 16.1 (7.9) | 19.9 (7.6)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Superiority; p < 0.001, ANCOVA

5. Secondary Outcome: Change in the 9 Hole Peg Test (9HPT) Score From Baseline
Description: 4 timed trials of the 9 hole peg test (9HPT) were performed and averaged (mean values are reported) for each separate hand (dominant and nondominant). The total time to complete the task is recorded for each trial and for each separate hand (dominant and nondominant). Longer times represent greater impairment.
Time Frame: Baseline - 2 weeks - 1 month - 3 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
seconds
  Baseline | 53.0 (24.3) | 52.2 (25.9)
  2 Weeks | 46.2 (21.3) | 53.4 (23.8)
  1 Month | 47.1 (21.9) | 55.8 (28.1)
  3 Months | 49.5 (20.5) | 54.2 (26.2)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Superiority; p < 0.001, ANCOVA

6. Secondary Outcome: Change in the 8-Meter Walking Time (8MW) Score From Baseline
Description: 4 timed trials of the 8 meter walking time (8MW) were performed and averaged (mean values are reported). Longer times represent greater impairment.
Time Frame: Baseline - 2 weeks - 1 month - 3 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
seconds
  Baseline | 9.4 (3.4) | 9.3 (3.3)
  2 Weeks | 8.0 (2.7) | 9.0 (3.9)
  1 Month | 7.8 (2.7) | 9.9 (5.0)
  3 Months | 8.4 (2.8) | 9.7 (4.1)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Superiority; p = 0.006, ANCOVA

7. Secondary Outcome: Change in Cerebellar Brain Inhibition (CBI) Measurements From Baseline
Description: Cerebellar brain inhibition (CBI) is expressed as motor evoked potential amplitude (average of 10 recordings). Lower values reflect higher inhibition and thus reduced impairment.
Time Frame: Baseline - 2 weeks - 1 month - 3 months
Measure: Mean (Standard Deviation); unit: millivolts
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 18 | 18
millivolts
  Baseline | 0.94 (0.12) | 0.88 (0.12)
  2 Weeks | 0.54 (0.13) | 0.91 (0.12)
  1 Month | 0.65 (0.14) | 0.95 (0.13)
  3 Months | 0.74 (0.11) | 0.90 (0.12)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Superiority; p < 0.001, ANCOVA

8. Secondary Outcome: Change in the Short-Form Health Survey 36 (SF36) Score From Baseline
Description: The Italian version of the Short-Form Health Survey 36 (SF-36): consists of 36 scaled score, yielding a total score of 0 (more disability) to 100 (less disability).
Time Frame: Baseline - 2 weeks - 1 month - 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 54.7 (17.5) | 55.3 (19.5)
  2 Weeks | 66.5 (17.5) | 57.9 (18.5)
  1 Month | 66.7 (16.8) | 60.1 (17.8)
  3 Months | 61.1 (18.8) | 56.3 (18.8)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Superiority; p = 0.043, ANCOVA

ADVERSE EVENTS:
Time Frame: 9 months
Description: Adverse event has been defined as any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Groups:
- Real tDCS, Then Sham tDCS: Participants who were randomized to receive real tDCS first and then sham tDCS
- Sham tDCS, Then Real tDCS: Participants who were randomized to receive sham tDCS first and then real tDCS
Arm/Group | Real tDCS, Then Sham tDCS | Sham tDCS, Then Real tDCS
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT03120013/Prot_SAP_000.pdf